CLINICAL TRIAL: NCT06855316
Title: Evaluating Combined Electromagnetic Stimulation for Enhanced Physical and Psychological Recovery in Athletes with DOMS: a Randomized Controlled Study
Brief Title: Evaluating Combined Electromagnetic Stimulation for Enhanced Physical and Psychological Recovery in Athletes with DOMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sierra Varona SL (Other)
Collaborators: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Alberto Sánchez Sierra, Director of Sierra Varona SL and professor at UCLM, Sierra Varona SL
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 017
Record Dates: First submitted 2025-02-05; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Recovery, Psychological; Transcranial Magnetic Stimulation
Keywords: transcraneal magnetic stimulation; delay onset muscle soreness; psychological profile

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: the outcome assessor will not know in which group is each participant, and the investigator will receive the data without knowing which data is from which group. Transcraneal magnetic stimulation in the placebo group was "applied"only with the sound reproduced by a speaker,remembering that the application of TMS is subthreshold, so the patient does not know if we are appying it or not, but all of them will here the same sound of the device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- control/placebo group (Placebo Comparator): Participants will be treated using the same device used in active stimulation groups, but the device will be turned off, thus providing a placebo effect. To maintain the placebo integrity, a pre-recorded sound mimicking the active device will be played during the session. Additionally, participants in the transcranial component will wear the machine's flap, similar to the TMS application, to further simulate the experience of active treatment. This method will ensure that the placebo control will be robust, allowing for accurate comparison with active treatments.
  Interventions: Device: electromagnetic stimulation
- Super Inductive (P) Group (Experimental): Participants in the Super Inductive (P) group will receivePeripheral Electromagnetic Stimulation (PES) following a Long-Term Potentiation (LTP) protocol. This protocol involved five cycles of stimulation at a frequency of 100 Hz, each lasting for 5 seconds, with a rest interval of 55 seconds between cycles. The total duration of the PES treatment will be approximately 10 minutes, as suggested by Lang et al. (2007) and Milanović et al. (2011) (Lang et al., 2007; Milanović et al., 2011). This stimulation aimes to enhance peripheral nerve activation and support recovery through localized neuromodulation.
  Interventions: Device: electromagnetic stimulation
- Transcranial (T) Group (Experimental): Participants in the Transcranial (T) group will get Transcranial Magnetic Stimulation (TMS) targeting at the primary motor cortex (M1). The protocol will be based on the findings of Dietmann et al. (2023) and Todd et al. (2003), consisting of the delivery of 2000 pulses of TMS over a minimum duration of 20 minutes (Dietmann et al., 2023; Todd et al., 2003). This intervention aimes to modulate cortical excitability, potentially enhancing muscle recovery through central nervous system adaptation.
  Interventions: Device: electromagnetic stimulation
- Combined Stimulation (Comb) Group (Experimental): Participants in the Combined (Comb) group will receive both TMS and PES simultaneously, providing a synergistic intervention aimed at optimizing recovery outcomes. The combined stimulation session will last 30 minutes, integrating the benefits of both central and peripheral modulation. This dual approach targets the M1 region for central effects while also stimulating peripheral nerves to promote localized recovery processes.
  Interventions: Device: electromagnetic stimulation

INTERVENTIONS:
Device: electromagnetic stimulation — After performing a high-intensity eccentric exercise session, participants will undergo a daily session of transcranial and/or peripheral magnetic stimulation for three days. The objective is to enhance nerve conduction, which, according to the latest theories on DOMS, may be the cause of decreased athletic performance

SUMMARY:
This randomized controlled trial explores the impact of a combined transcranial and peripheral electromagnetic stimulation over the potential correlation between psychological well-being and recovery outcomes of young athletes experiencing Delayed Onset Muscle Soreness.

DETAILED DESCRIPTION:
This randomized controlled trial explores the impact of a combined transcranial and peripheral electromagnetic stimulation (TMS and PES) over the potential correlation between psychological well-being and recovery outcomes of young athletes experiencing Delayed Onset Muscle Soreness. Grounded in the emerging theory of DOMS as an axonopathy affecting muscle spindles, this study examines whether paired-associative stimulation can show link over physical and psychological recovery processes. Forty-eight male athletes, aged 18 to 35 years, regularly engaged in exercise, will be randomly assigned to one of four groups: Control (placebo), PES, TMS, and Combined Stimulation (TMS + PES). All participants will perform a muscle-damaging exercise protocol to induce DOMS, followed by the assigned electromagnetic intervention. Assessments will include dynamometry, Counter Movement Jump (CMJ), Visual Analog Scale for Fatigue (VAS-F), Pain Pressure Threshold (PPT), sprint performance, and various psychological measures, such as the State-Trait Anxiety Inventory (STAI), Acceptance and Action Questionnaire-II (AAQ-II), and the Spanish versions of the Big Five Personality Traits, Perceived Stress Scale (PSS), and the Zung Self-Rating Depression Scale. These assessments will be conducted at baseline and at multiple intervals post-exercise (1 hour, 24 hours, 48 hours, and 72 hours).

ELIGIBILITY:
Inclusion Criteria:

1. be male,
2. aged between 18 and 35 years
3. engage in regular exercise at least three times per week for a minimum of one year
4. have no hypersensitivity to the areas designated for peripheral stimulation
5. be free from chronic conditions incompatible with exercise performance
6. have no recent musculoskeletal injuries to the lower limbs within the past six months,
7. be non-smokers
8. possess the cognitive capacity to understand the study's objectives and procedures.

Exclusion Criteria:

-

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-02-24 (Estimated); Primary Completion 2025-03-03 (Estimated); Study Completion 2025-03-07 (Estimated)

PRIMARY OUTCOMES:
Big Five Personality Trait Short Questionnaire (Spanish version) | Participants will complete questionnaires at 2 time points: just before treatment and after de last treatment (3 days after the first time frame).
  This tool is used to evaluate five core personality dimensions: neuroticism, extraversion, openness, agreeableness, and conscientiousness (Airagnes et al., 2021). The abbreviated version contains 10 items rated on a 5-point Likert scale, where 1 indicates "completely disagree" and 5 represents "completely agree." An example item from this questionnaire is, "I see myself as a person who gets nervous easily." This measure provided insight into the stable personality characteristics of the athletes and their potential impact on recovery and pain perception.Each item is rated on a Likert scale, typically ranging from 1 (Strongly Disagree) to 5 (Strongly Agree).
  Scores for each trait are summed up separately, with higher scores indicating stronger presence of that personality trait.
State-Trait Anxiety Inventory (STAI, Spanish version) | Participants will complete questionnaires at 2 time points: just before treatment and after de last treatment (3 days after the first time frame)
  To assess anxiety levels, the STAI will be used. Participants rated their responses on a 4-point Likert scale, where 1 means "not at all" and 4 means "very much," reflecting their state and trait anxiety. This measure allowed for an analysis of how anxiety levels might correlate with recovery outcomes and subjective pain experiences. It consists of 40 items, divided into two subscales:
  STAI-S (State Anxiety, 20 items): Assesses temporary feelings of anxiety in a specific moment.
  STAI-T (Trait Anxiety, 20 items): Measures a person's general tendency to experience anxiety over time.
  Each item is rated on a 4-point Likert scale:
  STAI-S: 1 (Not at all) to 4 (Very much so) STAI-T: 1 (Almost never) to 4 (Almost always) Scores range from 20 to 80 for each subscale, with higher scores indicating greater anxiety levels. The STAI is widely used in both clinical and research settings to assess anxiety in different populations.
Acceptance and Action Questionnaire-II (AAQ-II, Spanish version) | Participants will complete questionnaires at 2 time points: just before treatment and after de last treatment (3 days after the first time frame)
  The AAQ-II measures psychological inflexibility and experiential avoidance, which are critical in understanding how individuals cope with discomfort and stress (Carreira-Míguez et al., 2022). The 7-item questionnaire uses a 7-point Likert scale (0 = "never true" to 7 = "always true"), with higher scores indicating greater levels of psychological distress.The total score ranges from 7 to 49, with higher scores indicating greater experiential avoidance and psychological inflexibility, while lower scores reflect higher psychological flexibility. This scale is commonly used in clinical and research settings to evaluate mental health and intervention outcomes.
UCLA Loneliness Scale (Spanish version): | Participants will complete questionnaires at 2 time points: just before treatment and after de last treatment (3 days after the first time frame)
  The Spanish version of the Three-Item Loneliness Scale will be administered to assess perceived social isolation. Participants rated each of the three items on a 3-point scale, with 1 meaning "never" and 3 meaning "frequently." This scale helped to explore the role of social support and perceived isolation in recovery from physical exertion.The scale consists of 20 items, each rated on a 4-point Likert scale:
  1. (Never)
  2. (Rarely)
  3. (Sometimes)
  4. (Often) The total score ranges from 20 to 80, with higher scores indicating greater levels of loneliness. There is no strict cutoff, but higher scores generally reflect more significant perceived loneliness.
Zung Self-Rating Depression Scale (Spanish version): | Participants will complete questionnaires at 2 time points: just before treatment and after de last treatment (3 days after the first time frame)
  This self-applied scale contains 20 items designed to assess the severity of depressive symptoms, with both positive and negative formulations. The Zung scale's high specificity (over 80%) makes it a reliable tool for evaluating depression levels in the study's population (Carreira-Míguez et al., 2022). These baseline psychological assessments enabled the researchers to correlate psychological variables with recovery markers throughout the study.t consists of 20 questions, each evaluating various aspects of depression, including mood, physical symptoms, and psychomotor activity.
  Scoring
  Each question is rated on a 4-point Likert scale:
  1. (A little of the time)
  2. (Some of the time)
  3. (Good part of the time)
  4. (Most of the time)
  The total score ranges from 20 to 80, with higher scores indicating more severe depression:
  20-44: Normal range 45-59: Mild depression 60-69: Moderate to marked depression 70-80: Severe depression

CONTACTS AND LOCATIONS:
Locations (1):
- Alberto Sanchez Sierra, Toledo, TOLEDO, Spain

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: after publication during one year.